CLINICAL TRIAL: NCT07356167
Title: Passive Neurosensory Reintegration Training as a Tool to Augment Mild Traumatic Brain Injury
Acronym: PNRT for mTBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Erin Williams, Research Assistant Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20250973
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Mild Traumatic Brain Injury
Keywords: mTBI; mild traumatic brain injury; TBI; visuo-vestibular dysfunction; vestibular dysfunction
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive Neurosensory Reintegration Training (PNRT) (Experimental): Participants will receive Passive Neurosensory Reintegration Training (PNRT), a multisensory neuromodulation protocol integrating synchronized visual, vestibular, auditory, and somatosensory inputs to promote sensory reintegration and recovery of balance and oculomotor function. Each participant will complete 12 sessions over approximately two weeks (Days 1-12). Each session lasts approximately 60 minutes and involves exposure to coordinated low-intensity light, motion, and auditory stimuli in a controlled seated position. Participants will complete standardized assessments at Baseline, Day 6 (midpoint), Day 13 (post-intervention), and Day 40 (follow-up).
  Interventions: Device: Passive neurosensory reintegration training (PNRT)
- No Intervention - Controls (No Intervention): Participants assigned to the control arm will receive no active intervention during the initial 13-day period. They will undergo the same schedule of baseline, midpoint (Day 6), post (Day 13), and follow-up (Day 40) assessments as the PNRT group.

INTERVENTIONS:
Device: Passive neurosensory reintegration training (PNRT) — PNRT is a non-invasive, device-based system that delivers synchronized visual, vestibular, auditory, and somatosensory stimulation. The system consists of a light box and motion platform. Participants remain supine while receiving filtered halogen light at <10 lux intensity (non-laser, non-UV) synchronized with controlled stimuli.
  Arms: Passive Neurosensory Reintegration Training (PNRT)

SUMMARY:
Mild traumatic brain injury (mTBI) poses a substantial clinical and public health burden, often leading to persistent neurosensory and cognitive symptoms for which diagnostic and therapeutic solutions remain limited. This study proposes a multimodal diagnostic framework that integrates established mTBI screening tools and clinical neuro-optometric assessments with high-resolution oculomotor, vestibular, and reaction time (OVRT) testing to enhance diagnostic precision and identify prognostic markers of recovery. Normative data will be established in healthy controls to inform objective thresholds and support clinical implementation. Concurrently, we will evaluate the safety, tolerability, and preliminary efficacy of a novel, minimal-risk multisensory therapeutic intervention (i.e., passive neurosensory reintegration training, or PNRT) for individuals with sub-acute or chronic mTBI. By addressing critical gaps in both diagnosis and treatment, this project will improve mTBI recovery outcomes, inform future clinical trials, and advance evidence-based mTBI care guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 or older
2. Clear mechanism of injury (i.e., direct or indirect impact to head), or Any individual presenting with complaints of sudden (<24h) onset neurosensory symptoms as characterized by hearing a noise, feeling a force, or having an unexpected neurosensory perception and unexplained by any other known etiology ("sudden neurosensory events" or SNEs)
3. Glasgow Coma Scale (GCS) score of 13-15 at the time of injury
4. Observed or reported focal signs at the time of injury (e.g., loss of consciousness, amnesia, or confusion) or neurosensory symptoms (e.g., dizziness, headaches, photo/phonophobia, fatigue, vision problems, sleep changes, mood changes, cognitive fog) lasting over 4 weeks to 3 months (sub-acute), or over 3 months (chronic) following brain injury

Exclusion Criteria:

1. Any of the following: moderate to severe TBI characterized by penetrating head trauma, GCS <13 at the time of injury, LOC >30 minutes or PTA >24 hours, subdural or epidural hemorrhage for most recent occurence
2. mTBI/SNE Group: History of 4 or more clinically diagnosed mTBIs that warranted emergent assessment in a hospital or emergency department setting Control Group: History of mTBI within the last 12 months or presence of mTBI-related symptoms at time of enrollment
3. Presence of severe aphasia
4. History of diagnosed psychiatric disorder or autoimmune/rheumatologic conditions prior to brain injury

   1. Uncontrolled autoimmune/rheumatologic conditions including but not limited to Lyme, POTS, EDS, long COVID
   2. Psychiatric disorders: including but not limited to severe depression, schizophrenia, lupus)
5. Documented neurological disorders (e.g., epilepsy, stroke, dementia)
6. Legally blind (characterized by a best-corrected visual acuity of 20/200 or less in the better eye or a visual field of 20 degrees or less)
7. History of tumor of the brain or central nervous system
8. Actively receiving vision therapy for current mTBI-related visual-impairment
9. Wards of the state or prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Dizziness Handicap Inventory (DHI) Total Score | Baseline to Day 13 (Post-Intervention)
  Within-subject change in DHI total score from baseline to Day 13 following Passive Neurosensory Reintegration Training (PNRT). The mean change will be reported with 95% confidence intervals. Additionally, the proportion of participants achieving ≥18-point reduction in DHI score will be calculated as having clinically meaningful improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami Miller School of Medicine - Don Soffer Clinical Research Building, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in publications may be made available to qualified researchers upon reasonable request, following publication of primary study results.